CLINICAL TRIAL: NCT03853707
Title: A Phase I/IB Study of Ipatasertib in Combination With Carboplatin, Carboplatin/Paclitaxel, or Capecitabine/Atezolizumab in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Ipatasertib in Combination With Carboplatin, Carboplatin/Paclitaxel, or Capecitabine/Atezolizumab in Treating Patients With Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18496; NCI-2019-00465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18496 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2019-02-01; First posted 2019-02-26 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; Capecitabine; Carboplatin; ipatasertib; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (ipatasertib, carboplatin, paclitaxel) (Experimental): Patients receive ipatasertib PO QD on days 1-28. Patients also receive carboplatin IV over 30 minutes and paclitaxel IV over 60 minutes on days 1, 8, and 15 or days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Ipatasertib; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (ipatasertib and carboplatin) (Active Comparator): Patients receive ipatasertib PO QD on days 1-28. Patients also receive carboplatin IV over 30 minutes on days 1, 8, and 15 or days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Ipatasertib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm C (ipatasertib, capecitabine, atezolizumab) (Experimental): Patients receive ipatasertib PO QD on days 1-21, capecitabine PO BID on days 1-7 and 15-21, and atezolizumab IV over 30-60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Capecitabine; Drug: Ipatasertib; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
  Arms: Arm C (ipatasertib, capecitabine, atezolizumab)
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm C (ipatasertib, capecitabine, atezolizumab)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm A (ipatasertib, carboplatin, paclitaxel); Arm B (ipatasertib and carboplatin)
Drug: Ipatasertib — Given PO
  Other Names: GDC-0068; RG-7440
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm A (ipatasertib, carboplatin, paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies best dose of ipatasertib and how well it works with carboplatin with or without paclitaxel in treating patients with triple negative breast cancer that has spread to other places in the body (metastatic). Ipatasertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, paclitaxel, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving ipatasertib in combination with carboplatin, carboplatin/paclitaxel, or capecitabine/atezolizumab will work better in treating patients with triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) of ipatasertib plus carboplatin/paclitaxel (arm A), ipatasertib plus carboplatin (arm B), and ipatasertib, atezolizumab, and capecitabine (arm C) in patients with metastatic triple negative breast cancer (TNBC). (Phase I) II. To obtain initial evidence of activity by examining progression free survival for each dose regimen. (Phase IB)

SECONDARY OBJECTIVES:

I. To confirm the recommended phase II dose (RPIID) safety in expanded cohort by evaluating toxicities and confirm tolerability of the combinations.

II. To obtain evidence of activity by examining response rate based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

III. To evaluate clinical benefit rate (CBR), event-free survival, time-to-treatment failure and overall survival.

IV. Further describe the cumulative toxicities (Common Terminology Criteria for Adverse Events [CTCAE] 5.0) of the combinations.

V. To evaluate patient's quality of life (QOL).

EXPLORATORY OBJECTIVES:

I. To evaluate the progression-free survival and overall survival, based on the genomic alterations including PIK3CA/AKT/PTEN alterations and BRCA status.

II. To study the association of TNBC messenger ribonucleic acid (mRNA) expression profiling including Vanderbilt molecular subtype and treatment response.

III. To study the association of stool microbiome, calprotectin with diarrhea. IV. To study peripheral blood circulating tumor deoxyribonucleic acid (DNA). V. To study therapy resistance by analyzing tumor genomics and transcriptome analysis.

VI. To study the profiles of peripheral blood mononuclear cells and its association with response to therapy.

VII. To study genomic immune biomarkers and its association with response.

OUTLINE: This is a phase I, dose-escalation trial of ipatasertib, followed by a phase II trial. Patients are randomized or assigned to 1 of 3 arms depending on available slots.

ARM A: Patients receive ipatasertib orally (PO) once daily (QD) on days 1-28. Patients also receive carboplatin intravenously (IV) over 30 minutes and paclitaxel IV over 60 minutes on days 1, 8, and 15 or days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive ipatasertib PO QD on days 1-28. Patients also receive carboplatin IV over 30 minutes on days 1, 8, and 15 or days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive ipatasertib PO QD on days 1-21, capecitabine PO twice daily (BID) on days 1-7 and 15-21, and atezolizumab IV over 30-60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Ability to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically confirmed triple negative breast cancer defined by estrogen receptor (ER) or progesterone receptor (PR) =< 10% by immunohistochemistry (IHC) and HER2 negative defined by current American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guideline
* Disease progression during or following treatment with 0-2 lines of chemotherapy and/or biological targeted therapy in the metastatic setting
* Measurable (Arm C only) or non-measurable (allowed for Arm A or B) but evaluable disease per RECIST version (v)1.1 (Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation.)
* Baseline tissue requirement:

  * A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 20 x 5 um slides containing unstained, freshly cut, serial sections must be collected along with an associated pathology report prior to study enrollment
  * If only 10-19 slides are available, the patient may still be eligible for the study, after principal investigator approval has been obtained
  * If archival tumor tissue is unavailable or is determined to be unsuitable for required testing, tumor tissue must be obtained from a biopsy performed at screening
  * A biopsy may also be performed at screening if a patient's archival tissue test results do not meet eligibility criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1,500/uL) without granulocyte colony-stimulating factor support (obtained within 14 days prior to initiation of study treatment)
* Platelet count >= 100 x 10^9/L (100,000/uL) without transfusion (obtained within 14 days prior to initiation of study treatment)
* Hemoglobin >= 9 mg/dL (9 mg/dL) (patients may be transfused to meet this criterion) (obtained within 14 days prior to initiation of study treatment)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) (obtained within 14 days prior to initiation of study treatment), with the following exception:

  * Patients with documented liver or bone metastases may have AST and ALT =< 5 x ULN
* Alkaline phosphatase (ALP) =< 2 x ULN (obtained within 14 days prior to initiation of study treatment), with the following exceptions:

  * Patients with known liver involvement may have ALP =< 5 x ULN
  * Patients with known bone involvement may have ALP =< 7 x upper limit (UL)
* Serum bilirubin =< 1.5 x ULN (obtained within 14 days prior to initiation of study treatment) with the following exception:

  * Patients with known Gilbert disease: serum bilirubin level =< 3 x ULN
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 50 mL/min (calculated using the Cockcroft-Gault formula) (obtained within 14 days prior to initiation of study treatment)
* Partial thromboplastin time (PTT) (or activated partial thromboplastin time [aPTT]) and international normalized ratio (INR) =< 1.5 x ULN (except for patients receiving anticoagulation therapy) (obtained within 14 days prior to initiation of study treatment)
* Patients receiving heparin treatment should have a PTT (or aPTT) between 1.5 and 2.5 x ULN (or patient value before starting heparin treatment). Patients receiving coumarin derivatives should have an INR between 2.0 and 3.0 assessed in two consecutive measurements 1 to 4 days apart
* Fasting total glucose =< 150 mg/dL (obtained within 14 days prior to initiation of study treatment)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of study treatment. Women must refrain from donating eggs during this same period.

  * A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone- releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 6 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* Inability to comply with study and follow-up procedures
* >= grade 3 toxicities from previous treatment, not recovered to =< grade 2 at study entry
* Prior exposure to PI3K/AKT/mTOR pathway inhibitors including but not limited to everolimus, ipatasertib, gedatolisib or alpelisib etc
* Prior exposure to carboplatin for treatment of metastatic TNBC not allowed; prior treatment of carboplatin as neoadjuvant or adjuvant therapy allowed if last dose of therapy completed >= 12 months prior to initiation of the current study
* Prior exposure to paclitaxel or nab-paclitaxel for treatment of metastatic TNBC not allowed for carboplatin/paclitaxel arm; prior treatment of paclitaxel or nab-paclitaxel as neoadjuvant or adjuvant therapy allowed if last dose of therapy completed >= 12 months prior to initiation of the current study
* Prior exposure to capecitabine for treatment of metastatic TNBC not allowed for Arm C; prior treatment of capecitabine as adjuvant therapy allowed if the last dose of therapy completed >= 12 months prior to initiation of the current study for Arm C
* Prior treatment with immune check point inhibitors for Arm C
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment for Arm C
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions for Arm C:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor confirmation has been obtained
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* Active autoimmune disorders requiring steroid dose higher than prednisone 10 mg daily for Arm C
* Active disease or receiving treatment for hepatitis B or C or human immunodeficiency virus (HIV) infection for Arm C
* Receipt of a live, attenuated vaccine within 4 weeks prior to enrollment (start of treatment), during treatment, or within 5 months following the last dose of atezolizumab for Arm C
* Known allergy or hypersensitivity to any component of carboplatin and/or paclitaxel or nab-paclitaxel, or capecitabine (5-FU) formulation (for patients planned for the respective arms)
* Known dihydropyrimidine dehydrogenase (DPD) deficiency in patients selected to receive capecitabine for Arm C
* Known severe allergic reactions to cisplatin or other platinum-containing compounds or mannitol (for patients planned for platinum-containing arms)
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills
* Active infection requiring systemic anti-microbial treatment (including antibiotics, anti-fungals, and anti-viral agents)
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Known untreated or unstable brain metastasis or leptomeningeal metastasis from metastatic breast cancer
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  * Patients with indwelling catheters (e.g., PleurX) are allowed
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL, or corrected calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Known HIV infection
* Known clinically significant history of liver disease consistent with Child-Pugh class B or C, including active viral or other hepatitis (e.g., positive for hepatitis B surface antigen [HBsAg] or hepatitis C virus [HCV] antibody at screening), current drug or alcohol abuse, or cirrhosis

  * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV deoxyribonucleic acid [DNA] test) are eligible
  * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Prior allogeneic stem cell or solid organ transplantation
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of cycle 1 or anticipation of need for a major surgical procedure during the course of the study

  * Placement of a vascular access device is not considered major surgery
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 28 days after the last dose of ipatasertib, 5 months after the last dose of atezolizumab, and within 6 months after the last dose of paclitaxel, whichever occurs later

  * Women of childbearing potential (who are not postmenopausal with >= 12 months of non-therapy induced amenorrhea nor surgically sterile) must have a negative serum pregnancy test result either within 96 hours prior to day 1 of cycle 1 treatment
* New York Heart Association class II, III, or IV heart failure; left ventricular ejection fraction < 50%; or active ventricular arrhythmia requiring medication
* Current unstable angina or history of myocardial infarction within 6 months prior to day 1 of cycle 1 and cerebrovascular accident within 3 months prior to day 1 of cycle 1
* Congenital long QT syndrome or screening QT interval corrected using Fridericia's formula (QTcF) > 480 milliseconds
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion (including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction)
* Need for chronic corticosteroid therapy of >= 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease
* Treatment with approved or investigational cancer therapy within 14 days prior to day 1 of cycle 1
* Patients with a prior diagnosis of malignancy except non-melanomatous skin cancer treated >= 5 years ago are eligible, provided that they have not received prior taxanes or carboplatin as part of their prior treatment regimen, and that they meet all eligibility criteria
* Any other disease, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Yuan Y, Yost SE, Cui Y, Ruel C, Murga M, Tang A, Martinez N, Schmolze D, Waisman J, Patel N, Vora L, Tumyan L, Bozoghlanian M, Stewart D, Frankel PH. Phase I Trial of Ipatasertib Plus Carboplatin, Carboplatin/Paclitaxel, or Capecitabine and Atezolizumab in Metastatic Triple-Negative Breast Cancer. Oncologist. 2023 Jul 5;28(7):e498-e507. doi: 10.1093/oncolo/oyad026. PMID 37023705

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Ipatasertib, Carboplatin, Paclitaxel): Patients receive 300 mg ipatasertib PO QD on days 1-28. Patients also receive AUC 2 carboplatin IV over 30 minutes and 80 mg/m2 paclitaxel IV over 60 minutes on days 1, 8, and 15 or days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Ipatasertib and Carboplatin): Patients receive 300 mg ipatasertib PO QD on days 1-28. Patients also receive AUC 2 carboplatin IV over 30 minutes on days 1, 8, and 15 or days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm C (Ipatasertib, Capecitabine, Atezolizumab): Patients receive 300 mg ipatasertib PO QD on days 1-21, 750 mg/m2 capecitabine PO BID on days 1-7 and 15-21, and 840 mg atezolizumab IV over 30-60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab)
Started | 10 | 12 | 6
Completed | 10 | 12 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab) | Total
Number analyzed (Participants) | 10 | 12 | 6 | 28
Age, Continuous [Median (Full Range); unit: years] | 54 [49 to 75] | 54 [31 to 66] | 53 [48 to 60] | 53 [31 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 6 | 28
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2 | 1 | 1 | 4
  Asian | 1 | 1 | 0 | 2
  Hispanic | 1 | 6 | 3 | 10
  Non-Hispanic White | 6 | 4 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Estimated using the product-limit method of Kaplan and Meier. Failure defined as disease progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab)
Number analyzed (Participants) | 10 | 12 | 6
Months | 4.8 [2.8 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 3.9 [2.8 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 8.2 [4.6 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Secondary Outcome: Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab)
Number analyzed (Participants) | 10 | 12 | 6
Participants | 7 | 2 | 3

3. Secondary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial response (PR): At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR; Stable disease (SD): Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD; Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). Clinical Benefit Rate (CBR) = CR + PR + SD at 6 months.
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab)
Number analyzed (Participants) | 10 | 12 | 6
percentage of participants | 20.0 | 41.7 | 50.0

4. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the product-limit method of Kaplan and Meier. Failure defined as death from any cause.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab)
Number analyzed (Participants) | 10 | 12 | 6
Months | 11.2 [7.2 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 17.0 [9.5 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [11.1 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 3 years and 1 month.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm A (Ipatasertib, Carboplatin, Paclitaxel) | Arm B (Ipatasertib and Carboplatin) | Arm C (Ipatasertib, Capecitabine, Atezolizumab)
All-Cause Mortality (participants affected / at risk) | 6/10 | 10/12 | 1/6
Serious Adverse Events (participants affected / at risk) | 2/10 | 4/12 | 1/6
Other Adverse Events (participants affected / at risk) | 10/10 | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ipatasertib, Carboplatin, Paclitaxel) (N=10) | Arm B (Ipatasertib and Carboplatin) (N=12) | Arm C (Ipatasertib, Capecitabine, Atezolizumab) (N=6)
Fever (General disorders) | 0 (0) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ipatasertib, Carboplatin, Paclitaxel) (N=10) | Arm B (Ipatasertib and Carboplatin) (N=12) | Arm C (Ipatasertib, Capecitabine, Atezolizumab) (N=6)
Anemia (Blood and lymphatic system disorders) | 9 (43) | 9 (39) | 2 (15)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (7) | 5 (12) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (4) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (4)
Blurred vision (Eye disorders) | 2 (2) | 2 (5) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VISION CHANGES (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
darkening of vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (8) | 5 (12) | 1 (5)
Constipation (Gastrointestinal disorders) | 7 (12) | 10 (20) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 9 (51) | 12 (60) | 4 (25)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (10) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth Sore (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (5) | 2 (9) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (21) | 9 (37) | 5 (27)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oral sensitivity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (8) | 0 (0) | 0 (0)
Tooth broke off (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (9) | 6 (9) | 2 (6)
heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
mouth sore (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
oral sensitivity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
scratchy throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
tongue sensitivity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1)
Death NOS (General disorders) | 4 (4) | 10 (10) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 2 (12) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (17) | 10 (41) | 6 (49)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (12)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (15) | 0 (0)
Pain (General disorders) | 2 (3) | 6 (12) | 2 (5)
RIGHT BIG TOENAIL (General disorders) | 0 (0) | 1 (1) | 0 (0)
RIGHT BIG TOENAIL DISFGURED (General disorders) | 0 (0) | 1 (1) | 0 (0)
RIGHT BIG TOENAIL DISFIGURED (General disorders) | 0 (0) | 1 (11) | 0 (0)
RIGHT BIG TOENIAL DISFIGURED (General disorders) | 0 (0) | 1 (2) | 0 (0)
night sweats (General disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Right finger with pus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
AMAYLASE INCREASE (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (7) | 3 (8) | 3 (14)
Alkaline phosphatase increased (Investigations) | 4 (13) | 5 (11) | 4 (11)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 3 (8) | 4 (15)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 6 (10) | 5 (13) | 2 (15)
Creatinine increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (12) | 6 (20) | 3 (10)
Neutrophil count decreased (Investigations) | 10 (49) | 7 (47) | 2 (8)
Platelet count decreased (Investigations) | 1 (5) | 8 (35) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 9 (43) | 10 (60) | 4 (23)
Anorexia (Metabolism and nutrition disorders) | 4 (11) | 1 (1) | 4 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (7) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (9) | 9 (42) | 4 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (5) | 3 (20) | 3 (16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (11) | 3 (6) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (17) | 2 (4) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3) | 3 (11) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 5 (11) | 5 (17) | 2 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (25) | 7 (29) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (11) | 9 (23) | 2 (18)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (7) | 4 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (8) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 7 (28) | 1 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1) | 1 (6)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (7) | 2 (3)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 2 (6)
Dysgeusia (Nervous system disorders) | 2 (5) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 5 (21) | 2 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (28) | 6 (30) | 3 (18)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
brain fog (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (10)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (5) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (3)
Bleeding of old radiation burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 4 (11) | 2 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (9) | 2 (2)
SKIN PEELING (FINGERTIPS) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (6)
Flushing (Vascular disorders) | 2 (2) | 4 (7) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (3) | 1 (11)
Hypertension (Vascular disorders) | 9 (46) | 10 (47) | 4 (29)
Hypotension (Vascular disorders) | 3 (5) | 3 (8) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03853707/Prot_SAP_000.pdf